CLINICAL TRIAL: NCT02235168
Title: Effect of Rollator on Walking Distance in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Doctor in Physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 6MWTElderly
Record Dates: First submitted 2014-08-25; First posted 2014-09-09 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- With rollator (Experimental): Six minutes walking test with rollator
  Interventions: Procedure: six minute walking test
- Without rolator (Active Comparator): Six minutes walking test without rollator
  Interventions: Procedure: six minute walking test

INTERVENTIONS:
Procedure: six minute walking test

SUMMARY:
To evaluate the effect of a rollator on 6 Minute Walking Test (6MWT) in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* elderly people (older than 60 years)

Exclusion Criteria:

* respiratory diseases

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
six minute walking test | 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium